CLINICAL TRIAL: NCT07315815
Title: Physiological Effects of Controlled vs. Assisted Ventilation During Moderate-to-severe Acute Respiratory Distress Syndrome (PEARL Study)
Brief Title: Physiological Effects of Controlled vs. Assisted Ventilation During Moderate-to-severe ARDS (PEARL Study)
Acronym: PEARL
Status: Not yet recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, BELLO GIUSEPPE, Principal Investigator, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 7648
Record Dates: First submitted 2025-12-18; First posted 2026-01-02 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2025-11

CONDITIONS: Ventilator-Induced Lung Injury
MeSH Terms: conditions — Ventilator-Induced Lung Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Background:

In patients with acute hypoxemic respiratory failure or ARDS, mechanical ventilation is often required. Two common strategies are pressure support ventilation (PSV), which allows spontaneous breathing, and volume-controlled ventilation (VCV), which delivers fixed tidal volumes. Although PSV can improve comfort, strong inspiratory efforts may cause excessive lung inflation and increase the risk of ventilator-induced lung injury (VILI). In contrast, VCV with muscle paralysis ensures full control over tidal volume and driving pressure, potentially offering better lung protection.

Hypothesis:

The study will help determine whether a controlled ventilation strategy - with or without volume adjustments and with or without muscle paralysis - provides superior lung protection compared to PSV in hypoxemic patients with intense inspiratory effort.

Methods:

This prospective physiological study will be performed in the ICU of Fondazione Policlinico Universitario A. Gemelli (Rome, Italy) and will include 20 moderate to severe ARDS patients. Each patient will undergo four 30-minute ventilation phases:

PSV with clinical PEEP;

VCV at 6 ml/kg predicted body weight (PBW);

VCV with muscle paralysis and Vt equal to PSV;

VCV with muscle paralysis and Vt adjusted to keep driving pressure ≤14 cmH₂O.

During each phase, data on gas exchange, respiratory mechanics, inspiratory effort, and regional ventilation (via electrical impedance tomography) will be collected.

Endpoints:

Primary: Regional tidal volume distribution during VCV vs. PSV.

Secondary: Transpulmonary driving pressure, dorsal ventilation fraction, and pendelluft occurrence.

Expected Impact:

By comparing assisted and controlled ventilation under different conditions, the study aims to clarify which strategy better balances patient comfort, effective ventilation, and lung protection in ARDS patients with high respiratory drive.

DETAILED DESCRIPTION:
This is a prospective, single center, physiological interventional study designed to investigate the respiratory mechanics and regional lung ventilation effects of assisted versus fully controlled mechanical ventilation in patients with moderate to severe acute respiratory distress syndrome (ARDS). The study is conducted in a tertiary care intensive care unit and focuses on short term physiological responses to different ventilatory strategies under controlled experimental conditions. The study specifically evaluates how ventilation mode and tidal volume targeting influence regional lung inflation, inspiratory effort, and risk of ventilator induced lung injury using advanced physiological monitoring tools, including esophageal pressure measurement and electrical impedance tomography.

The scientific rationale is based on the observation that assisted ventilation modes, such as pressure support ventilation, preserve spontaneous breathing but may expose patients with high respiratory drive to excessive tidal volumes and transpulmonary pressures. This condition is associated with patient self inflicted lung injury and regional lung overdistension. Fully controlled ventilation allows strict control of tidal volume and driving pressure and may reduce regional lung stress and strain. However, direct physiological comparison between assisted and controlled ventilation under standardized conditions remains limited. This study evaluates whether switching patients with high inspiratory effort to volume controlled ventilation, either maintaining tidal volume observed during assisted ventilation or targeting protective driving pressure values, improves regional ventilation homogeneity and reduces markers of lung overdistension while preserving gas exchange.

After enrollment, patients undergo four sequential ventilatory phases applied in a fixed order. Each phase lasts 30 minutes. The first 25 minutes allow physiological stabilization and adaptation to the ventilatory mode. The final 5 minutes are used for signal acquisition and physiological measurements. The four phases include assisted ventilation with clinically selected pressure support and positive end expiratory pressure, volume controlled ventilation targeting 6 ml per kg predicted body weight, volume controlled ventilation with tidal volume matched to tidal volume measured during assisted ventilation with neuromuscular blockade, and volume controlled ventilation targeting 6 ml per kg predicted body weight with neuromuscular blockade and driving pressure titration to remain at or below 14 cmH2O. During neuromuscular blockade phases, respiratory rate is adjusted based on arterial blood gas analysis to maintain physiological pH and PaCO2 targets.

Respiratory mechanics are assessed using combined airway, esophageal, and gastric pressure measurements obtained through a balloon catheter nasogastric tube system. Flow and airway pressure are measured using a pneumotachograph. Signals are acquired digitally and stored for offline analysis. Derived parameters include inspiratory effort, transpulmonary pressure swings, respiratory system and lung driving pressure, lung and chest wall compliance, respiratory muscle activity, pressure time product, and occlusion pressure indices. Static respiratory mechanics are assessed using standardized inspiratory and expiratory occlusion maneuvers. These measurements allow detailed characterization of patient ventilator interaction, lung stress, and mechanical energy transfer to the respiratory system.

Regional ventilation distribution is assessed using electrical impedance tomography. A dedicated electrode belt positioned at the mid thoracic level continuously records impedance changes at high temporal resolution. Offline analysis includes calculation of tidal ventilation distribution between dependent and nondependent lung regions, estimation of regional tidal volume, ventilation homogeneity indices, pixel level ventilation heterogeneity, end expiratory lung impedance changes, and detection of pendelluft phenomenon. Recruitment volume is estimated by comparing end expiratory impedance at different positive end expiratory pressure levels. These measurements provide high resolution functional imaging of regional lung aeration and ventilation distribution during each ventilatory phase.

Physiological and gas exchange parameters collected during each phase include tidal volume, respiratory rate, airway pressures, arterial blood gases, and work of breathing indices. Data acquisition is standardized across all study phases to ensure comparability between ventilatory strategies.

The study follows a physiological repeated measures design. Continuous variables are summarized using median and interquartile range. Categorical variables are expressed as proportions. Due to the small sample size and expected non normal distribution of physiological variables, non parametric statistical tests are used. Global comparisons across study phases are performed using the Friedman test. Pairwise comparisons are performed using Wilcoxon signed rank test or McNemar test when appropriate. Statistical significance is defined using two sided p values less than or equal to 0.05. Statistical analyses are performed using validated statistical software.

Because of the physiological exploratory design and absence of prior data describing regional lung inflation behavior under identical experimental conditions, formal power calculation was not performed. The planned enrollment target is 20 patients. This sample size is consistent with previous physiological crossover studies investigating respiratory mechanics and regional lung ventilation using advanced monitoring techniques. The selected sample size is considered sufficient to detect clinically meaningful physiological differences between ventilation strategies and to generate hypothesis generating data for future clinical outcome trials.

Safety monitoring is performed throughout the study. All adverse events occurring during study procedures are recorded. Adverse events related to medical devices are classified according to applicable European medical device regulations. Incidents, device deficiencies, and serious incidents are reported to the competent national authority and device manufacturer according to regulatory requirements. Serious incidents include events leading to death, serious deterioration in health status, or serious public health risk. Device related safety monitoring includes assessment of device performance, reliability, and usability during study procedures.

Data are collected using standardized data collection tools and stored in secure institutional systems. Raw physiological waveforms are stored for offline analysis. Data quality is ensured through predefined acquisition protocols, standardized measurement procedures, and centralized offline analysis performed by trained investigators. Physiological signals undergo quality review before analysis to ensure signal integrity and measurement accuracy.

The study is planned over a 12 month enrollment period. Follow up data include hospital survival status recorded after completion of study procedures. The study is conducted according to institutional clinical research standards and applicable regulatory requirements for interventional physiological studies.

ELIGIBILITY:
Inclusion Criteria:

* Intubated patients fulfilling moderate-to-severe ARDS (ratio of arterial partial pressure of oxygen to fraction of inspired oxygen.
* Undergoing assisted ventilation as per clinical decision

Exclusion Criteria:

* refusal to participate, age younger than 18 years old, pregnancy
* contraindication to EIT use (e.g., presence of pacemaker or automatic implantable cardioverter defibrillator), impossibility to place the EIT belt in the right position (e.g., presence of surgical wounds dressing), and any contraindication to the insertion of a nasogastric tube (e.g., recent upper-gastrointestinal surgery, esophageal varices).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Intubated patients fulfilling ARDS criteria and undergoing assisted ventilation as per clinical decision will be enrolled in case of moderate-to-severe hypoxemia.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Regional tidal volume during volume-controlled vs. pressure support ventilation | 1 year

IPD SHARING:
Plan to Share IPD: No